CLINICAL TRIAL: NCT03761329
Title: A Randomized Controlled Trial to Investigate the Efficacy of a Bier's Block Compared to a Mini-bier's Block in Patients Undergoing Hand Surgery
Brief Title: Bier's Block Versus Mini-bier's Block in Patients Undergoing Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18.46/ANESTH18.03
Record Dates: First submitted 2018-10-16; First posted 2018-12-03 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Surgery; Anesthesia, Local
Keywords: Anesthesia; Bier's block; Mini-Bier's block; Hand surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bier's block (Active Comparator): Upperarm intravenous regional anesthesia (Bier's block) with lidocaine 0.5% 40ml
  Interventions: Procedure: Conventional Bier's block with lidocaine 0.5% 40ml
- Mini-Bier's block (Experimental): Forearm intravenous regional anesthesia (mini-Bier's block) with lidocaine 0.5% 25ml
  Interventions: Procedure: mini-Bier's block with lidocaine 0.5% 25ml

INTERVENTIONS:
Procedure: mini-Bier's block with lidocaine 0.5% 25ml — An intravenous catheter will be placed in the dorsal vein of the hand that will undergo surgery. Afterwards, a tourniquet will be placed on the forearm and inflated, after which the anesthetic can be administered via the dorsal vein catheter (25ml lidocaine 0.5%). The tourniquet remains inflated for 10 minutes to reduce systemic toxicity reactions postoperatively.
  Other Names: forearm intravenous regional anesthesia (IVRA)
  Arms: Mini-Bier's block
Procedure: Conventional Bier's block with lidocaine 0.5% 40ml — An intravenous catheter will be placed in the dorsal vein of the hand that will undergo surgery. Afterwards, a tourniquet will be placed on the upper arm and inflated, after which the anesthetic can be administered via the dorsal vein catheter (40ml Lidocaine 0.5%). The tourniquet remains inflated for 25 minutes to reduce systemic toxicity reactions postoperatively.
  Other Names: Upperarm intravenous regional anesthesia (IVRA)
  Arms: Bier's block

SUMMARY:
By means of an observer-blinded, randomized controlled trial, the analgesic efficacy of an upper-arm Bier's block and a forearm mini-Bier's block will be investigated in patients undergoing hand surgery. The hypothesis is that there is no difference between the two types of anesthetic techniques with respect to the analgesic efficacy.

DETAILED DESCRIPTION:
Introduction:

Several ways of anesthesia can be used to perform hand surgery, being general anesthesia, intravenous regional anesthesia as well as locoregional anesthesia. Locoregional anesthesia and intravenous regional anesthesia are often performed since patients can be discharged from the hospital more rapidly.

A conventional Bier's block is performed using a tourniquet on the upper arm to create a bloodless field and to contain the anesthetics within the surgical area (1). Complications are rare but are often linked to a systemic toxicity reaction after releasing the tourniquet (2). A mini-Bier's block in which the tourniquet is placed on the fore-arm, has been shown to be a safe and effective way of anesthesia to perform hand surgery. By using this type of anesthesia, the dose of the anesthetic can be reduced compared to a conventional Bier's block which reduces the risk of systemic toxicity reactions (3-5).

Currently, studies that made a comparison between the two anesthesia techniques are scarce and inconsistent. Next to that, those studies also used different types of anesthetics and dosages. To see which technique is advantageous in clinical practice, the investigators want to investigate the efficacy of the Bier's block and mini-Bier's block in patients that are planned to undergo hand surgery.

Outcome measures:

The primary aim of this study is to compare the analgesic efficacy of the Bier's block versus the mini-Bier's block. The hypothesis is that there is no difference between the two techniques. A blinded surgeon will determine the analgesic efficacy of these techniques (graded as "complete" or "incomplete") and divide the efficacy in 4 grades. Grade 1 and grade 2 are considered "complete" blockade, while grade 3 and grade 4 are considered "incomplete" blockade. Grade 1: complete motor and sensory blockade, grade 2: partial motor blockade but no pain or deep pressure sensitivity, grade 3: partial motor blockade with mild pain requiring rescue local or opioid analgesia, grade 4: incomplete motor- and sensory blockade requiring sedation/conversion to general anesthesia).

Secondary study outcomes:

* Onset time, which is defined as the time from the injection of the local anesthetic until the complete sensory loss in hand (assessed by the blinded surgeon via "pin prick").
* Patient's pre-, intra- and post-operative pain scores will be measured via an 11-point Numeric Rating Scale (NRS) in which number 0 means "no pain at all", number 5 means "moderate pain" and number 10 means "worst possible pain".
* Tourniquet time: the amount of time that the tourniquet is inflated.
* Tourniquet tolerance time: the amount of time required for the inflated tourniquet to cause a painful sensation (NRS > 3).
* Satisfaction with the surgical field (bloodless field) will be graded by a blinded surgeon, measured using a 5-point scale (1= extremely dissatisfied until 5= extremely satisfied).
* The time spent in the operating room.
* Duration of surgery.
* General patient satisfaction will be assessed using a 7-point Likert Scale, in which number 1 equals "extremely dissatisfied" and number 7 means "extremely satisfied".

Design:

In this monocentric, investigator-initiated, observer-blinded, prospective, randomized, controlled, non-inferiority trial, 2 anaesthetic procedures will be compared in patients that undergo hand surgery (Carpal Tunnel Syndrome, trigger finger, dequervain tenovaginitis, disease of Dupuytren, ganglion cyst).

This study will be performed according to the Declaration of Helsinki and will be approved by the ethics committee of the JESSA Hospital, Hasselt, Belgium before the start of the study. A written informed consent will be obtained before participation in the study.

Randomization will be performed using a computer-generated random allocation sequence. Allocation numbers will be sealed in opaque envelopes, which will be opened in sequence by an independent anesthesiologist who is not involved in the assessment of outcomes.

Both the surgeon and the researcher will be blinded for the used type of anesthesia. Since the clear difference between an upper arm and forearm tourniquet, all patients will receive a second tourniquet which will not be inflated. That is, patients receiving the Bier's block will receive an additional forearm tourniquet which will not be inflated and patients in group of the mini-Bier's block will receive an additional upperarm tourniquet which will not be inflated. In this way, a possible de-blinding of the surgeon and researcher is minimized.

Study Procedures:

The patient will first receive information about this study. Before the start of the study, written informed consent will be obtained, after which the patient will be randomized to one of the 2 treatment groups. Before surgery, all patients will receive an intravenous catheter in the contralateral arm with infusion of 0.9% Natriumchloride (NaCl), paracetamol 1g and standard monitoring (non-invasive blood pressure, electrocardiogram and O2 saturation measurements).

In the Bier's block group:

An intravenous catheter will be placed in the dorsal vein of the hand that will undergo surgery. Afterwards, a tourniquet will be placed on the upper arm and inflated, after which the anesthetic can be administered via the dorsal vein catheter (40ml Lidocaine 0.5%). The tourniquet remains inflated for 25 minutes to reduce systemic toxicity reactions postoperatively.

In the mini-Bier's block group:

An intravenous catheter will be placed in the dorsal vein of the hand that will undergo surgery. Afterwards, a tourniquet will be placed on the forearm and inflated, after which the anesthetic can be administered via the dorsal vein catheter (25ml lidocaine 0.5%). The tourniquet remains inflated for 10 minutes to reduce systemic toxicity reactions postoperatively.

Before the start of the surgery, the blinded surgeon will assess the quality of the block (primary outcome) using a forceps. The quality of the block will be graded "complete" or "incomplete" as described above. In case of grade 1 or grade 2, the surgical procedure can start. In case of grade 3, the blockade will be enhanced (local anesthetic or intravenous opioid administration (alfentanil or sufentanil)). In case of grade 4, sedation/conversion to general anesthesia will be performed.

All secondary outcome measures will be investigated by the blinded researcher.

Statistical analysis:

Sample size was determined for the primary study outcome with the aim to reject the non-inferiority of the mini-Bier's block. Based on a meta-analysis (unpublished data) we expect a 98.5% complete blockade in the experimental group (mini-Bier's block) and a 100% complete blockade in the control group (Bier's block). With a difference of 5% between the 2 groups and a binary outcome (complete/incomplete), we calculated that 135 patients are needed per group (α=0.05, power=0.80). Considering a drop-out rate of 3.5%, the total number of patients is 140 per group.

Descriptive statistics will be presented as frequencies and percentages of the total amount of patients for categorical variables, while numerical variables will be presented as mean. Group comparison will be performed using Chi-square test (or a Fisher's Exact test when necessary) for frequencies. Depending on normality, a Mann-Whitney U test or a Student's t-test will be used. Corrections will be applied for multiple measurements of the Numerical Rating Scale (NRS) for pain scores. An average difference of 1.3 points or more on the NRS pain score is considered clinical relevant. A p-value <0.05 is considered statistical significant, while p<0.10 is considered a tendency.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* American Society of Anesthesiology (ASA) physical status classification: 1-3
* Patients planned to undergo hand surgery which can be performed using either a Bier's block or a mini-Bier's block

Exclusion Criteria:

* < 18 years old
* Patients that participate in other clinical, pharmaceutical trials or trials with medical devices
* Patients that previously have been randomized in this trial
* Patients that need to undergo surgery using sedation/general anesthesia
* Bilateral surgery
* BMI ≥ 40 kg/m2
* History of neurological conditions
* Chronic pain symptoms
* Concomitant use of Opioids in the last month
* Diabetes mellitus with organ damage
* Oversensitivity to local anesthetics
* Blood clotting disorders
* Inability to understand and adhere to the study design

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Sensory and motor block of the hand | 5 minutes after injection of lidocaine 0.5%
  This study wants to evaluate and compare the analgesic efficacy of the Bier's block with the mini-Bier's block. The blinded surgeon will assess the analgesic effectivity and grade it as either complete (grade 1 and grade 2) or incomplete (grade 3 and grade 4). Grade 1 is defined as complete motor and sensory blockade; grade 2 is defined as partial motor blockade with no pain or deep pressure sensitivity. Grade 3 is defined as partial motor blockade with mild pain and the need for rescue local or opioid analgesia. Grade 4 is defined as incomplete motor and sensory blockade requiring sedation/conversion to general anesthesia.

SECONDARY OUTCOMES:
Pre-operative pain score: Numeric Rating Scale (NRS) | Before the start of anesthesia technique
  Pain score before the start of anesthesia technique (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Pain due to anesthesia technique: Numeric Rating Scale (NRS) | At the end of performing the anesthesia technique
  Pain caused by performing the anesthesia technique (measured via an 11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Tourniquet time | From start of inflation until deflation of the tourniquet
  Total time the tourniquet is inflated
Onset time of analgesia | At injection of the anaesthetic until complete blockade of the sensory nerves
  Onset time of analgesia (starts at injection of the anaesthetic and will continue until complete blockade of the sensory nerves (assessed via pin prick)). When after 10 minutes no sensory blockade occurred, rescue medication (alfentanil (0,5 mg)) will be applied. When alfentanil (0,5 mg) will not provide enough sensory blockade, sedation with diprivan (titration per 1cc) or, if required, conversion to general anesthesia will be applied.
Tourniquet tolerance time | From start of inflation until deflation of the tourniquet
  Time required for the tourniquet to cause a painful sensation (NRS > 3)
Pain score at start of surgery (surgical incision): Numeric Rating Scale (NRS) | At the start of the surgical procedure
  Pain score at surgical incision (start of surgical procedure) (11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable)
Satisfaction with surgical conditions (bloodless field) assessed by the surgeon with a 5-point likert scale | At the start of the surgical procedure
  Satisfaction with surgical conditions (bloodless field): assessed by the surgeon with a 5-point scale. This scale is ranged (1, 2, 3, 4, 5) in which 1 stands for "completely dissatisfied" and 5 for "completely satisfied".
Intraoperative pain score: Numeric Rating Scale (NRS) | every 5 min during the surgical procedure
  Pain score (11-point Numeric Rating Scale where 0 = no pain and 10 is worst pain imaginable) at every 5 min during the surgical procedure (both surgical pain and tourniquet pain)
Time in operating room | From entering the operating room until leaving the operating room
  Time the patient is in operating room (start by entering the operating room until leaving the operating room)
Time of surgical procedure | From start of surgical incision until closing of the surgical wound
  Time of surgical procedure (start at surgical incision until closing of the surgical wound)
General satisfaction of the patient: Likert scale | Assessed on day 1 post surgery
  General satisfaction of the patient with the anesthesia technique (measured via a 7-point Likert scale, with 1 being completely dissatisfied and 7 being completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stessel, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiao FB, Chen J, Lesser JB, Resta-Flarer F, Bennett H. Single-cuff forearm tourniquet in intravenous regional anaesthesia results in less pain and fewer sedation requirements than upper arm tourniquet. Br J Anaesth. 2013 Aug;111(2):271-5. doi: 10.1093/bja/aet032. Epub 2013 Mar 18. PMID 23508563
- [Background] Guay J. Adverse events associated with intravenous regional anesthesia (Bier block): a systematic review of complications. J Clin Anesth. 2009 Dec;21(8):585-94. doi: 10.1016/j.jclinane.2009.01.015. PMID 20122591
- [Background] Arslanian B, Mehrzad R, Kramer T, Kim DC. Forearm Bier block: a new regional anesthetic technique for upper extremity surgery. Ann Plast Surg. 2014 Aug;73(2):156-7. doi: 10.1097/SAP.0b013e318276da4c. PMID 23407261
- [Background] Karalezli N, Karalezli K, Iltar S, Cimen O, Aydogan N. Results of intravenous regional anaesthesia with distal forearm application. Acta Orthop Belg. 2004 Oct;70(5):401-5. PMID 15587026
- [Background] Chong AK, Tan DM, Ooi BS, Mahadevan M, Lim AY, Lim BH. Comparison of forearm and conventional Bier's blocks for manipulation and reduction of distal radius fractures. J Hand Surg Eur Vol. 2007 Feb;32(1):57-9. doi: 10.1016/j.jhsb.2006.10.002. Epub 2006 Nov 22. PMID 17123673